CLINICAL TRIAL: NCT01185639
Title: Phase II Study of Stereotactic Body Radiation Therapy (SBRT) After First-Line Chemotherapy for Metastatic NSCLC
Brief Title: Stereotactic Body Radiation Therapy (SBRT) in Metastatic Non-small Cell Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00013994; NCI-2010-01877 (Registry Identifier: CTRP); CCCWFU 62110 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2010-08-18; First posted 2010-08-20 (Estimated); Results first posted 2019-11-29 (Actual); Last update posted 2019-11-29 (Actual); Status verified 2019-11

CONDITIONS: Non-Small-Cell Lung Carcinoma; Liver Cancer; Adrenal Cancer
Keywords: lung cancer; metastatic; SBRT; Stereotactic body radiation therapy; liver; spine; adrenal; bone cancer; Spinal Column
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Liver Neoplasms; Adrenal Gland Neoplasms; Lung Neoplasms; Neoplasm Metastasis; Bone Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- SBRT for metastatic NSCLC (Experimental): SBRT for lung lesions, liver lesions, adrenal lesions, spinal lesions
  Interventions: Radiation: stereotactic body radiation therapy

INTERVENTIONS:
Radiation: stereotactic body radiation therapy — For lung, liver, axial skeleton, and adrenal tumors a dose of either 54 Gy in 3 fxs or 5000 cGy in 5 fx using SBRT techniques
  Other Names: Elekta Bodyframe; Cyberknife

SUMMARY:
This protocol is a single arm phase II multi-center trial evaluating the efficacy of Stereotactic Body Radiation Therapy (SBRT) in patients with oligometastatic non-small cell lung cancer (NSCLC) with response or stable disease after 4 cycles of first-line chemotherapy. The core hypothesis tested is that SBRT after 4 cycles of first-line chemotherapy is feasible, safe, provides durable local control of treated lesions and improves time to progression compared to historical controls. Patients are eligible for enrollment if they have metastatic NSCLC with ≤5 lesions amenable to SBRT.

ELIGIBILITY:
Inclusion Criteria:

General

* Patients with AJCC sixth edition metastatic non-small cell lung carcinoma
* Pathologic diagnosis of stage 4 non-small cell lung cancer prior to enrollment.
* Patients must have response or stable disease by RECIST criteria after 4 cycles of first-line chemotherapy
* Maximum of number of lesions per patient will be 5 total. .
* Patients with solitary brain metastases previously treated with surgery or stereotactic radiosurgery (+/- WBRT) and currently controlled at the time of study enrollment are also eligible. Patients with history of brain metastases must have an MRI showing no active brain metastases within 80 days of study enrollment. Patients with a history of brain metastases may have up to 5 extracranial sites of disease except for those with an untreated primary tumor where section 3.1.3.3 will also apply.
* Patients with newly diagnosed stage IV NSCLC with an untreated primary must no more than 3 active extracranial metastatic lesions other than the primary site and regional lymph nodes.
* Age ≥ 18 years old
* Performance Status 0-2 (ECOG)
* A signed study specific consent form is required.

Lung (only applies to patients with active lung lesions)

* Patients cannot have more than 3 lung lesions
* Local failure after surgical resection will be consider a metastatic lesion for purposes of protocol inclusion.
* All lung lesions must be visible on CT imaging
* Cumulative diameter of lung lesions must be <7cm
* Patients may have active mediastinal disease in a single mediastinal nodal station if he/she has not received prior mediastinal RT
* Must meet criteria regarding status of primary tumor site described in section 3.1.9.
* Must be able to anticipate achieving SBRT dosimetry guidelines
* Must have adequate lung function defined within 90 days of enrollment as: (1) Forced Expiratory Volume in 1 second (FEV1) >30% of predicted or >800 Ml, (2) diffusing capacity of the lung for carbon monoxide (DLCO) >30 % predicted and (3) no evidence of actively worsening respiratory status

Liver (only applies to patients with active liver lesions

* Patients cannot have more than 3 liver lesions
* All active liver lesions must be discrete on CT or MRI imaging
* Combined diameter of all liver lesions must be <6cm
* Must be able to anticipate achieving SBRT plan per dosimetry guidelines for the liver.
* Liver function tests (AST, ALT, total bilirubin) should be within ≤ 3 times the upper limit of normal (ULN)
* Serum Albumin must be >2.5g/dL
* Patients cannot have active ascites.

Adrenal Gland

* Unilateral adrenal disease
* Must be able to anticipate achieving the SBRT plan per dosimetry guidelines.

Bone Lesions

* Treatment of any bone lesion is permissible if it is anticipated that the dosimetry guidelines can be met.

Spine and Paraspinal lesions

* Patients cannot have more than 3 vertebrae or paraspinal sites involved (each involved vertebral body or paraspinal site is scored as 1 site of disease)
* Must be no clinical or radiographic evidence of spinal cord compression
* If spinal metastases is within previously irradiated field, there must be a 6 month interval between prior radiation course and study enrollment
* Prior spinal cord maximum dose at level of vertebral disease must be ≤50Gy

Exclusion Criteria:

* Primary tumor progression on first-line chemotherapy
* Patients with complete response to first-line chemotherapy with no measurable target for SBRT
* >5 metastatic lesions or >3 metastatic lesions in patients with an untreated primary site are ineligible (ipsilateral hilar and mediastinal lymph nodes are considered part of an untreated primary site and are not counted as metastatic lesions)
* Solitary brain metastases and an untreated node positive primary tumor, without other extracranial metastases amenable to SBRT are ineligible
* Retreatment of previously irradiated tumor will be excluded per 3.1.9.2 above.
* Mediastinal lymph nodes involving multiple mediastinal nodal stations or N3 disease are ineligible.
* Pleural effusion known to be malignant or visible of chest xray.
* Untreated brain metastases
* Bilateral adrenal metastases
* Metastases in other sites not considered amenable to SBRT
* Patients with liver metastases cannot have received prior upper abdominal radiation
* Prior radiation to spine (most commonly in treatment of primary lung cancer), cannot have received >50Gy to the spinal cord at the level of current vertebral metastases
* Clinical or radiographic evidence of spinal cord compression are ineligible
* Patients with serious, uncontrolled, concurrent infection(s).
* Weight loss (>10% of body weight) in the prior 3 months.
* Pregnant or lactating women

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2010-08 (Actual); Primary Completion 2016-06-27 (Actual); Study Completion 2016-06-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Blackstock, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (2):
- United States (2):
  - Coastal Carolina Radiation Oncology, Wilmington, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina

REFERENCES:
- [Derived] Petty WJ, Urbanic JJ, Ahmed T, Hughes R, Levine B, Rusthoven K, Papagikos M, Ruiz JR, Lally BE, Chan M, Clark H, D'Agostino RB Jr, Blackstock AW. Long-Term Outcomes of a Phase 2 Trial of Chemotherapy With Consolidative Radiation Therapy for Oligometastatic Non-Small Cell Lung Cancer. Int J Radiat Oncol Biol Phys. 2018 Nov 1;102(3):527-535. doi: 10.1016/j.ijrobp.2018.06.400. Epub 2018 Jul 10. PMID 30003996

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SBRT for Metastatic NSCLC
Started | 29
Completed | 27
Not Completed | 2
Not completed — Progressed and didn't receive therapy | 2

BASELINE CHARACTERISTICS:
Arm/Group | SBRT for Metastatic NSCLC
Number analyzed (Participants) | 27
Age, Continuous [Median (Full Range); unit: years] | 65 [49 to 83]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 26
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival
Description: Actuarial progression-free survival will be determined using the product-limit method of Kaplan and Meier and will be reported with an exact 95% confidence interval. Using the RECIST criteria including progression of the protocol treated tumors, non-protocol treated tumors and the development of new metastatic disease. Only protocol treated tumors will be determined by RECIST defined as complete lesion disappearance or <25%or original size; partial >30% decrease of target lesion; stable <30% decreased of target lesion and; local failure increase >20% of target lesion. Non-protocol tumor progression will be determined by the treating physician. Measured by imaging every 3 months.
Time Frame: up to 2 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | SBRT for Metastatic NSCLC
Number analyzed (Participants) | 27
months | 11.2 [7.6 to 15.9]

2. Secondary Outcome: To Assess Physical Function for This Cohort of Patients
Description: Using the Vulnerable Elders Survey (VES-13) A 13-item self-reporting questionnaire includes age, self-rated health, limitations in physical function and disability to assess for deterioration of physical function/health. Scoring for the VES-13 is as follows: Total scores are summed together based on self-rated health (0-1), physical function (0-2), functional disability (0-4), (range from 0 to 7). A total score of 3 or more identifies participants as vulnerable to the risk of decline of physical function.
Time Frame: up to 3 months after treatment
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | SBRT for Metastatic NSCLC
Number analyzed (Participants) | 27
Score on a scale | 2 (2.7)

3. Secondary Outcome: Number of Participants With Local Control
Description: Local control (LC) of SBRT-treated lesions will only be assessed in patients with at least 4-months of radiographic follow-up.
Time Frame: up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | SBRT for Metastatic NSCLC
Number analyzed (Participants) | 27
Participants | 1

4. Secondary Outcome: Overall Survival
Description: Overall survival will be reported with an exact 95% confidence interval.
Time Frame: up to 4 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | SBRT for Metastatic NSCLC
Number analyzed (Participants) | 27
months | 28.4 [14.5 to 45.8]

5. Secondary Outcome: Impact of Treatment on Quality of Life (FACT-L)
Description: Using the Functional Assessment of Cancer Therapy - Lung (FACT-L) a 36-item self-administered questionnaire evaluating physical, social/family, emotional, and functional well-being; subscales (symptoms, cognitive function, regret of smoking) on a five-point scale from 0 (not at all) to 4 (very much). Maximum score 136. Subscale scores added to obtain total score. The higher the score the greater the impact on the quality of life.
Time Frame: up to 3 months after treatment
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SBRT for Metastatic NSCLC
Number analyzed (Participants) | 27
score on a scale | 100.3 (23.7)

ADVERSE EVENTS:
Time Frame: 90 days following the end of radiation therapy will be recorded and graded on the AE Log. Only those toxicities Grade 3 and above will be reported.
Description: Only Grade 3 or higher adverse events that were possibly related to stereotactic body radiation therapy were collected for this study.
Arm/Group | SBRT for Metastatic NSCLC
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 0/27
Other Adverse Events (participants affected / at risk) | 1/27
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SBRT for Metastatic NSCLC (N=27)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) — Grade 2 related to stereotactic body radiation therapy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes